CLINICAL TRIAL: NCT00081900
Title: A Phase 1/2 Study of DENSPM (N1, N11-diethylnorspermine) in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: A Safety and Efficacy Study of DENSPM in Patients With Liver Cancer Who Are Not Eligible for Surgical Care
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated early by Genzyme because there were insufficient data to support clinical benefit to HCC patients on the study.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GD3-165-101
Record Dates: First submitted 2004-04-26; First posted 2004-04-28 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — N(1),N(11)-diethylnorspermine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DENSPM (Experimental)
  Interventions: Drug: DENSPM )

INTERVENTIONS:
Drug: DENSPM ) — Each patient will receive DENSPM at an initial dose of 30mg/m^2, then escalating to 120mg/m^2, single IV infusion on D1,3,5,8,10,12 of every 28 days as one cycle, planned for 8 cycles if no withdrawn occur
  Other Names: diethylnorspermine

SUMMARY:
Approximately 18-45 patients with Hepatocellular Carcinoma (HCC) will be treated with DENSPM at approximately 5 centers in the United States. First, we will be trying to determine the highest dose that can be given safely and is well tolerated (this is called the maximally tolerated dose, or the MTD, for short). Once that is established, we will enroll additional patients to learn more about potential side effects and to see whether DENSPM can slow the growth of HCC tumors. We also want to learn about the safety of DENSPM. Many medications used to treat cancer cause side effects (discomforts or illness). In this study, we want to understand what side effects occur in patients with HCC who are treated with DENSPM.Study was terminated after initial assessment of insufficient data to support clinical benefit in this population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven HCC, or if the patient is not a medically appropriate candidate for biopsy, then all of the following criteria must be met: A.History of cirrhosis or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV)infection. B.A focal liver lesion ≥ 3 cm on CT or MRI with arterial hypervascularization. C.Confirmation of the liver lesion by a second imaging modality (US/ CT/ MRI).D.AFP ≥1000 ng/ml, or ≥ 4000 ng/ml if Hepatitis B surface Ag positive.
* For recurrent HCC, radiographic evidence of progression.
* Not appropriate for curative therapy (surgical resection) or refuses potentially curative therapy
* Measurable disease, defined as having at least one measurable intrahepatic tumor lesion (using Response Criteria in Solid Tumors [RECIST]). Prior therapy is acceptable only if there is documented progression of the selected measurable lesion(s) following completion of the therapy.
* Required laboratory values
* Renal function: serum creatinine ≤1.2mg/dL Hematologic function: leukocyte count ≥1,500/mm3, platelet count ≥50,000/mm3 Hepatic function: transaminases ≤5x upper limit normal (ULN), albumin ≥2.0g/dL, total bilirubin ≤3.5mg/dL Sodium: ≥130mEq/L
* Karnofsky Performance Status of ≥ 60%
* CLIP Score ≤ 3
* If female and of childbearing potential, must use an effective method of contraception
* Willing and able to provide written informed consent

Exclusion Criteria:

* Has received localized therapy (e.g., radiotherapy, RFA, injection therapy, or chemoembolization)within 6 weeks prior to treatment, Day1. Prior local lesion-specific radiotherapy is acceptable only if the treated lesion(s) is/are not the only source of measurable disease or there is documented progression of the treated lesion(s) following completion of the therapy.
* Has received any other systemic therapy for HCC within 3 weeks prior to treatment, Day 1. Prior therapy is acceptable only if there is documented progression following completion of the therapy.
* Has received another investigational therapy within 30 days prior to study entry
* Has any unstable serious or life-threatening medical condition, other than HCC (e.g., unstable angina, other cancer diagnosis with the exception of basal cell carcinoma, or patients with prior malignancy except for adequately treated basal cell carcinoma(s), in situ cervical cancer, or other cancer for which the patient has been disease-free for five or more years)
* Newly noted clinically significant electrocardiogram (ECG) abnormality
* Clinically significant abnormal laboratory result that is not consistent with patient's clinical course
* Active gastrointestinal bleeding resulting in clinically significant hemodynamic changes or a reduction in hemoglobin.
* Active inflammatory bowel disease (IBD) and/or active gastric or duodenal ulcer disease
* Has a history of central nervous system (CNS) metastases, seizure disorder or neurological exam finding suggestive of CNS metastases
* Has Stage B or C liver cirrhosis according to Child-Pugh-Turcotte Classification
* Has ascites refractory to diuretic therapy
* Has any contraindication for MRI procedure
* If female of childbearing potential, has a positive serum HCG
* If female, is lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-03; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine the overall safety profile of DENSPM intravenous infusion in patients with unresectable HCC. | 8 months
To establish the MTD and dose limiting toxicities of DENSPM intravenous infusion in patients with unresectable HCC. | 8 months

SECONDARY OUTCOMES:
To evaluate antitumor response as measured by progression free survival when DENSPM is administered for up to eight 28 day cycles in patients with advanced HCC. | 8 months
To evaluate the pharmacokinetics of DENSPM in plasma and HCC tissue in patients unresectable HCC. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (8):
  - University of Illinois- Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Partners Cancer Care, Boston, Massachusetts
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - McGuire VA Medical Center, Richmond, Virginia